CLINICAL TRIAL: NCT05231941
Title: Comparison of Intraoperative Intravenous Lidocaine Infusion and Transversus Abdominis Plane (TAP) Block for Post-operative Analgesia Following Laproscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Haris Sheikh, Post-Graduate Trainee, Department of Anaesthesiology, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5515
Record Dates: First submitted 2022-01-19; First posted 2022-02-09 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine Group (Experimental): After induction of anaesthesia, a bolus of 2mg/kg intravenous lidocaine will be given followed by Lidocaine infusion at the rate of 1.5 mg/kg/hour which will be stopped at the end of surgery.
  Interventions: Drug: Lidocaine IV
- TAP group (Experimental): After completion of procedure and before extubation, bilateral ultrasound guided subcoastal transversus abdominis plane (TAP) block will be performed by the primary anaesthetist. After taking aseptic measures, with patient in supine position a high frequency (6-13 MHz) linear ultrasound probe will be placed obliquely just inferior to the costal margin over the anterior abdominal wall. With the help of a 21G or 22G, 100 mm needle, 20 ml of 0.375% Ropivacaine will be injected between rectus sheath and fascia of transversus abdominis muscle, bilaterally.
  Interventions: Drug: Ropivacaine
- Control group (No Intervention): No additional intervention will be given to this group

INTERVENTIONS:
Drug: Lidocaine IV — Bolus and infusion of lidocaine will be administered
  Arms: Lidocaine Group
Drug: Ropivacaine — Bilateral TAP block will be given to these patients
  Arms: TAP group

SUMMARY:
This study is aimed to determine the post operative pain after laparoscopic cholecystectomy by dividing patients into three different group. Group A will receive lidocaine 2mg/kg bolus at induction followed by 1.5mg/kg/hr infusion. Group B will receive bilateral subcostal TAP block with 0.375% 20ml Ropivicaine on each side. Group C will not receive any additional pain regime apart from the routine intraoperative analgesics. Pain score will be assessed post operatively for 24 hours at regular intervals using visual analog score.

ELIGIBILITY:
Inclusion Criteria:

* Age group (18-65)
* Undergoing elective Laproscopic Cholecystectomy
* ASA status I or II

Exclusion Criteria:

* Participation in any other trial
* Known hypersensitivity to study medications
* Chronic Opioid used
* Seizure disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Pain score | On arrival in PACU (0 hours)
  Pain score will be assessed using visual analog scoring system (0: No pain and 10: Worst Imaginable Pain)
Pain score | At 2 hours
  Pain score will be assessed using visual analog scoring system (0: No pain and 10: Worst Imaginable Pain)
Pain score | At 4 hours
  Pain score will be assessed using visual analog scoring system (0: No pain and 10: Worst Imaginable Pain)
Pain score | At 6 hours
  Pain score will be assessed using visual analog scoring system (0: No pain and 10: Worst Imaginable Pain)
Pain score | At 12 hours
  Pain score will be assessed using visual analog scoring system (0: No pain and 10: Worst Imaginable Pain)
Pain Score | At 24 hours
  Pain score will be assessed using visual analog scoring system (0: No pain and 10: Worst Imaginable Pain)

SECONDARY OUTCOMES:
Post operative nausea and vomiting | On arrival, At 2 hours, 4 hours, 6 hours, 12 hours and 24 hours
  Nausea and vomiting score would be assess using Bellville scoring system (0: No nausea or vomiting, 1: nausea, 2: nausea and belching, 3: vomiting)
Patient Satisfaction | At 24 hours or discharge
  Patient satisfaction will be assessed on Likert Scale (Completely Disagree, Disagree, Neutral, Agree, Completely Agree)

CONTACTS AND LOCATIONS:
Overall Officials: Haris Sheikh, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan